CLINICAL TRIAL: NCT00077428
Title: Phase II Trial of PS-341 (NSC 681239) Followed by the Addition of Doxorubicin at Progression in Advanced Adenoid Cystic Carcinoma of the Head and Neck
Brief Title: Bortezomib Followed by the Addition of Doxorubicin at Disease Progression in Treating Patients With Locally Advanced, Recurrent, or Metastatic Adenoid Cystic Carcinoma (Cancer) of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02574; E1303; U10CA021115 (NIH); CDR0000350319 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Salivary Gland Cancer; Salivary Gland Adenoid Cystic Carcinoma; Stage III Adenoid Cystic Carcinoma of the Oral Cavity; Stage III Salivary Gland Cancer; Stage IV Adenoid Cystic Carcinoma of the Oral Cavity; Stage IV Salivary Gland Cancer
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Bortezomib; Doxorubicin

ARMS (1):
- Treatment (bortezomib, doxorubicin hydrochloride) (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression continue to receive bortezomib as above and doxorubicin IV over 2-5 minutes on days 1 and 8. Treatment repeats every 21 days for up to 14 courses in the absence of further disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Drug: doxorubicin hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well bortezomib followed by doxorubicin at the time of disease progression works in treating patients with locally advanced, recurrent, or metastatic adenoid cystic carcinoma (cancer) of the head and neck. Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Drugs used in chemotherapy, such as doxorubicin, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining bortezomib with doxorubicin may kill more tumor cells

DETAILED DESCRIPTION:
OBJECTIVES: Primary I. Determine the objective tumor response in patients with locally advanced, recurrent, or metastatic adenoid cystic carcinoma of the head and neck treated with bortezomib.

Secondary I. Determine the time to progression in patients treated with this drug. II. Determine the overall survival of patients treated with this drug. III. Determine the toxic effects of this drug in these patients. IV. Determine the objective tumor response, time to progression, and overall survival of patients who progress on single-agent bortezomib and are then treated with doxorubicin and bortezomib.

V. Determine the toxic effects of this regimen in these patients. VI. Determine the profile and concentration of inflammatory and angiogenic cytokines in serum of patients before and in response to this regimen.

VII. Correlate the expression of biomarkers which may be affected by the ubiquitin-proteasome degradation pathway (NF-kB, p53, p27, cyclin D1, cyclin E, vascular endothelial growth factor [VEGF], MVD, V-CAM, and N-CAM) on tumor tissue with the clinical activity of bortezomib in these patients.

OUTLINE: This is a multicenter study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression continue to receive bortezomib as above and doxorubicin IV over 2-5 minutes on days 1 and 8. Treatment repeats every 21 days for up to 14 courses in the absence of further disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 8 years.

PROJECTED ACCRUAL: A total of 23-37 patients will be accrued for this study within 2.3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenoid cystic carcinoma of the head and neck

  * Locally advanced, recurrent, or metastatic disease that is considered incurable by known therapies
* Unidimensionally measurable disease
* Must not have stable disease for at least 9 months before study entry
* No known brain metastases
* Performance status - ECOG 0-2
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* AST and ALT no greater than 2.5 times upper limit of normal
* Bilirubin normal
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* LVEF at least lower limit of normal by MUGA
* No history of congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No active or ongoing infection
* No prior allergy to compounds of similar chemical or biological composition to bortezomib
* No other concurrent uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* No pre-existing neuropathy > grade 1
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* See Chemotherapy
* No prior anthracyclines, including any of the following:

  * Doxorubicin
  * Epirubicin
  * Daunorubicin
  * Idarubicin
* No prior mitoxantrone
* No prior high-dose chemotherapy for bone marrow transplantation
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* At least 3 weeks since prior radiotherapy
* At least 3 weeks since prior surgery
* More than 4 weeks since prior investigational drugs
* No other concurrent anticancer therapy or agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-06; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Objective tumor response (complete and partial overall response) as defined by Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 10 years

SECONDARY OUTCOMES:
Toxicities, based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 | Up to 30 days after last dose of study treatment
Progression free survival | Time from randomization or registration to the earlier of disease recurrence or death from any cause, assessed up to 10 years
  Examined using Kaplan-Meier estimates.
Overall survival | Time from randomization or registration to date of death (from any cause) or date of last contact, assessed up to 10 years
  Examined using Kaplan-Meier estimates.
Association of change in cytokine concentration with response to bortezomib therapy | Up to 1 hour post-treatment (course 2)
  A Wilcoxon rank sum test at a two-sided 10% significance level will be used
Correlation of the expression of biomarkers which may be affected by the ubiquitin-proteasome degradation pathway on tumor tissue with clinical activity | Baseline
  Estimated using Fisher's exact test at a two-sided 10% significance level.

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios Argiris, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States